CLINICAL TRIAL: NCT02122250
Title: Developing and Testing Accessible Web-based Support for Patient Self-management of Diabetes
Brief Title: Web-based Support for People With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 4746
Record Dates: First submitted 2013-03-21; First posted 2014-04-24 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Health literacy; web intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Interactive web-based materials (Experimental): Interactive web-based materials for self-management of diabetes
  Interventions: Behavioral: Interactive web-based materials
- Static web-based materials (Active Comparator): Static version of the interactive web-based materials
  Interventions: Behavioral: Static web-based materials

INTERVENTIONS:
Behavioral: Interactive web-based materials — Interactive web-based materials for self-management of diabetes
  Arms: Interactive web-based materials
Behavioral: Static web-based materials — Static web-based materials
  Arms: Static web-based materials

SUMMARY:
This project will address vital questions regarding how best to design web-based materials for the growing population of patients with basic literacy and computer skills but lower levels of health literacy, building on our previous experience of developing web-based materials for people with lower levels of literacy and health literacy.

This study will be carried out two phases. Phase 1 will use qualitative methods to understand user experiences of the web-based materials through observational 'think-aloud' interviews with users. Phase 2 will test the newly developed web-based materials to a static (non-interactive) version of the materials online.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants are patients with Type 2 diabetes aged 18 years or more, who are able to consent.

Exclusion Criteria:

* Severe mental health problems, palliative care, recent bereavement, known opposition to involvement in research or inability to complete research measures, e.g. learning disability, inability to read / speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1041 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
user engagement | This will be measured by intervention completion rates

SECONDARY OUTCOMES:
Patient enablement | Participants will be followed up as soon as they finished looking at the website, which is expected to be 20-40 minutes after they start the study.
Website satisfaction | Participants will be followed up as soon as they finished looking at the website, which is expected to be 20-40 minutes after they start the study.
Physical activity attitudes and intentions | Participants will be followed up as soon as they finished looking at the website, which is expected to be 20-40 minutes after they start the study.
Diabetes and Physical activity knowledge | Participants will be followed up as soon as they finished looking at the website, which is expected to be 20-40 minutes after they start the study.

OTHER OUTCOMES:
Single item: whether you would recommend the website to others | Participants will be followed up as soon as they finished looking at the website, which is expected to be 20-40 minutes after they start the study.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Yardley, Principal Investigator — University of Southampton